CLINICAL TRIAL: NCT02794207
Title: Home or Away From Home: Patient-Centered Outcomes Related to the Management of Neutropenia Which Are Most Important to Children With AML and Their Caregivers
Brief Title: Home or Away From Home - Descriptive Interviews (Aim 2)
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Primary Children's Hospital (Other); Texas Children's Cancer Center (Other); Children's Healthcare of Atlanta (Other); C.S. Mott Children's Hospital (Other); Children's Medical Center Dallas (Other); Arkansas Children's Hospital Research Institute (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); Children's Hospital of Michigan (Other); Lucile Packard Children's Hospital (Other); Seattle Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 15-012082
Record Dates: First submitted 2016-05-13; First posted 2016-06-09 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Pediatric Acute Myeloid Leukemia
Keywords: Pediatric; Cancer; AML; Qualitative Interview
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Participants: One qualitative, semi-structured interview will be conducted. Each interview will last approximately 30-45 minutes and may be audio recorded (if consent is provided). Interviews will consist of several open-ended questions focusing on having the participant reflect upon past experiences with neutropenia management and the impact of the participant's illness and treatment. Several close-ended questions regarding participant's thoughts on potential outcomes will also be included.
- Caregivers: One qualitative, semi-structured interview will be conducted. Each interview will last approximately 30-45 minutes and may be audio recorded (if consent is provided). Interviews will consist of several open-ended questions focusing on having the participant reflect upon past experiences with neutropenia management and the impact of their child's illness and treatment. Several close-ended questions regarding participant's thoughts on their child's potential outcomes will also be included.

SUMMARY:
The primary objectives of this study are to identify what outcomes related to the management of neutropenia are most important to children with AML and their caregivers. Patients who have completed treatment for AML and their caregivers will be interviewed in order to better understand the impact of neutropenia management on children with AML and their families. The primary outcome of these interviews is to identify patient-centered outcomes related to neutropenia management to include in a subsequent comparative-effectiveness analysis. Investigators will use these data to develop a structured survey for administration to prospectively identified patients in subsequent studies.

DETAILED DESCRIPTION:
Treatment for pediatric acute myeloid leukemia (AML) involves intensive chemotherapy regimens that result in periods of profound neutropenia leaving patients susceptible to severe infectious complications. There are little clinical data to inform whether management of neutropenia post AML chemotherapy should occur in an outpatient or inpatient setting. Further, no studies have been conducted that assess the impact of neutropenia management strategy on the quality of life of pediatric patients with AML. Given that infectious complications are the leading cause of treatment related mortality among AML patients, it is important to identify the neutropenia management strategy that will lead to the best clinician- and patient- identified outcomes in order to improve the care of these patients.

This is a qualitative interview study where interviews of patients and/or caregivers will be performed. Participants will be patients less than 19 years of age at diagnosis (and their caregivers) receiving or having received chemotherapy for AML from eleven participating pediatric hospitals across the United States. Participants (children and caregivers) will be interviewed in an effort to develop a survey that captures patient- and caregiver- identified outcomes related to neutropenia management.

ELIGIBILITY:
Inclusion Criteria:

1. To be enrolled in this study, patients must be:

   * A male or female between 8 and 22 years of age
   * Have a diagnosis of AML
   * Be either within 6-12 months of completion of the second course of chemotherapy for AML OR out of AML therapy for up to 3 years
2. To be enrolled in this study, caregivers must be:

   * A male or female 18 years of age or older
   * Be the parent/legal guardian of a child that meets the inclusion criteria detailed above (#1) OR
   * Be the parent/legal guardian of a male or female child younger than 8 years of age with AML and who is within 6-12 months of completion of their second course of chemotherapy
   * Be the parent/legal guardian of a male or female child younger than 8 years of age with AML and who is out of AML therapy for up to 3 years
3. Parental/guardian informed consent and, if appropriate, child assent.

Exclusion Criteria:

1) None

Ages: 8 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Study population will consist of patients who are less than 19 years of age at the time of diagnosis (and their caregivers) receiving or having received chemotherapy for AML.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-01-03 (Actual); Study Completion 2017-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Aplenc, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (11):
- United States (11):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Lucile Packard Children's Hospital, Palo Alto, California
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Children's Hospital of Michigan, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Medical Center of Dallas, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Only aggregate level data will be shared with the study sponsor Patient-Centered Outcomes Research Institute (PCORI).

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participants | Caregivers
Started | 32 | 54
Completed | 32 | 54
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data werenot collected for caregivers.
Groups:
- Patients: Patients who participated in a qualitative interview about their experience with AML. One qualitative, semi-structured interview was conducted. Each interview lasted approximately 30-45 minutes and may be audio recorded (if consent is provided).
- Caregivers: Caregivers who participated in a qualitative interview about their experience with AML. One qualitative, semi-structured interview was conducted. Each interview lasted approximately 30-45 minutes and may be audio recorded (if consent is provided).
- Total: Total of all reporting groups
Arm/Group | Patients | Caregivers | Total
Number analyzed (Participants) | 32 | 0 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23 |  | 23
  Between 18 and 65 years | 9 |  | 9
  >=65 years | 0 |  | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.4 (6.54) |  | 14.4 (6.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 |  | 17
  Male | 15 |  | 15
Region of Enrollment [Number; unit: participants]
  United States | 32 |  | 32

OUTCOME MEASURES:

1. Primary Outcome: Issues Related to Type of Neutropenia Management That Are Most Important to Children and Their Caregivers.
Description: Issues related to type of neutropenia management are not quantifiable. All interviewees gave unique responses to issues related to neutropenia management, and themes were identified after all interviews were conducted and analyzed.
Time Frame: One qualitative semi-structured interview was conducted post-neutropenia management. The interview lasted about 30-45 minutes.
Population: All participants (patients and caregivers) who participated in the semi-structured interviews. 3 key, novel themes were identified across these interviews.
Measure: Number; unit: key themes identified
Groups:
- Participants: One qualitative, semi-structured interview will be conducted. Each interview lasted approximately 30-45 minutes and were audio recorded (if consent is provided). Interviews consisted of several open-ended questions focusing on having the participant reflect upon past experiences with neutropenia management and the impact of the participant's illness and treatment. Several close-ended questions regarding participant's thoughts on potential outcomes were also included.
Arm/Group | Participants
Number analyzed (Participants) | 86
key themes identified | 3

ADVERSE EVENTS:
Time Frame: Adverse events were not collected while interviews were being conducted. Interviews were conducted when a patient was within 6-12 months of the completion of their second course of chemotherapy or up to 3 years out following the completion of all their frontline AML chemotherapy. The time relative to treatment, therefore, varied by family.
Description: There is no study intervention; this is a qualitative interview study only, thus adverse events were a non-issue and not monitored or assessed.
Arm/Group | Participants | Caregivers
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No